CLINICAL TRIAL: NCT06411561
Title: A Multi-Modal Combination Intervention to Promote Cognitive Function in Older Intensive Care Unit Survivors
Acronym: SLEEP-COG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Maya Elias, PhD, RN, Assistant Professor, School of Nursing, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00018228; K23AG078448 (NIH)
Record Dates: First submitted 2024-04-11; First posted 2024-05-13 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Critical Illness; Delirium; Cognitive Impairment; Cognitive Decline; Alzheimer's Disease; Dementia; Circadian Dysrhythmia; Sleep Disturbance
MeSH Terms: conditions — Critical Illness; Delirium; Cognitive Dysfunction; Alzheimer Disease; Dementia; Parasomnias | interventions — Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SLEEP + COG (Experimental): * Combination of SLEEP and COG interventions, for up to 7 days/nights + usual post-ICU inpatient care
  * Personalized timing of morning, afternoon, or evening COG sessions, based on CSM scale at baseline
  Interventions: Behavioral: SLEEP + COG
- COG (Experimental): * Daily 30-minute computerized cognitive training sessions (Lumosity), for up to 7 days + usual post-ICU inpatient care
  * Personalized timing of morning, afternoon, or evening COG intervention sessions, based on CSM scale at baseline
  Interventions: Behavioral: COG
- SLEEP (Experimental): - Nighttime use of earplugs and eye masks, for up to 7 nights + usual post-ICU inpatient care
  Interventions: Behavioral: SLEEP
- AC (Active Comparator): - Active comparator condition; delivery of educational modules on brain health + usual post-ICU inpatient care
  Interventions: Behavioral: AC

INTERVENTIONS:
Behavioral: SLEEP + COG — Combination of SLEEP and COG interventions
  Arms: SLEEP + COG
Behavioral: COG — Daily 30-minute session of computerized cognitive training
  Arms: COG
Behavioral: SLEEP — Nighttime use of both ear plugs and eye masks
  Arms: SLEEP
Behavioral: AC — Educational modules on cognitive and sleep health
  Arms: AC

SUMMARY:
Up to 25% of intensive care unit (ICU) survivors experience cognitive impairment comparable in severity to mild Alzheimer's disease and related dementias after hospital discharge. Older ICU survivors (ages 60 and older) are at highest risk for delirium and subsequent cognitive impairment, which contribute to higher risk for cognitive decline related to Alzheimer's disease and related dementias. Sleep and activity are essential for recovery from critical illness, yet ICU survivors experience both sleep deficiency and profound inactivity. About 75-80% of ICU patients experience circadian dysrhythmia, which contributes to cognitive decline and increases likelihood of developing Alzheimer's disease and related dementias. The scientific premises of the proposed study are: 1) a combined sleep promotion and cognitive training intervention will have synergistic effects to mitigate the risk of cognitive impairment and development of Alzheimer's disease and related dementias in older ICU survivors; and 2) chronotherapeutic timing of interventions (i.e., adjusting timing of interventions according to circadian rhythm) may improve intervention efficacy.

DETAILED DESCRIPTION:
Using a 2 x 2 factorial design, 100 English- or Spanish-speaking older ICU survivors will be enrolled after discharge out of ICU and randomized to one of 4 combinations of two interventions: SLEEP and COG. We propose that the combination of a nighttime sleep promotion intervention [SLEEP: nighttime use of earplugs and eye masks] and a daytime computerized cognitive training intervention [COG: daily 30-minute cognitive training sessions] may produce synergistic effects on cognitive function to mitigate delirium and reduce risk of incident Alzheimer's disease and related dementias. Because circadian dysrhythmia contributes to cognitive decline, chronotherapeutic timing of the COG intervention could maximize intervention efficacy.

Specific Aim 1: Test the separate and combined effects of SLEEP and COG [SLEEP + COG, SLEEP, COG] versus an active control [AC] in improving cognitive function for older ICU survivors.

Specific Aim 2: Examine circadian rhythm parameters of continuous body temperature (iButton: wearable sensor) to determine the optimal window for timing of the COG intervention.

Specific Aim 3: Examine if the effects of each intervention on cognitive function are mediated by sleep and activity, and examine if selected biological and clinical factors moderate intervention effects.

Exploratory Aim 4: Explore the effect of each intervention on cognitive function at 1 month and incident Alzheimer's disease and related dementias at 6 months and 12 months post-hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 60 years old
* Current hospitalization at University of Washington Medical Center or Harborview Medical Center
* Intensive care unit (ICU) length of stay greater than 24 hours
* Recovery from critical care status to acute care status, and/or discharge out of ICU
* Fluent in English or Spanish
* Functional independence on activities of daily living prior to hospitalization (Katz Index = 6)

Exclusion Criteria:

* Documented history or suspicion of Alzheimer's disease or dementia, or current prescription of anti-dementia medication
* Documented history of bipolar disorder or schizophrenia
* Documented acute stroke or traumatic brain injury
* Severe vision impairment
* Severe hearing impairment
* Severe paralysis or dominant arm paresis
* Transfer from skilled nursing care facility or inpatient rehabilitation facility

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | Post-intervention/within 7 days of hospital discharge
  RBANS Update: Repeatable Battery for the Assessment of Neuropsychological Status; total index score, range: 40-160; higher scores indicate better performance
Cognitive function | Follow-up at 1 month post-hospital discharge
  RBANS Update: Repeatable Battery for the Assessment of Neuropsychological Status; total index score, range: 40-160; higher scores indicate better performance
Cognitive function | Follow-up at 6 months post-hospital discharge
  RBANS Update: Repeatable Battery for the Assessment of Neuropsychological Status; total index score, range: 40-160; higher scores indicate better performance
Cognitive function | Follow-up at 12 months post-hospital discharge
  RBANS Update: Repeatable Battery for the Assessment of Neuropsychological Status; total index score, range: 40-160; higher scores indicate better performance

SECONDARY OUTCOMES:
Cognitive function: executive function, working memory | Post-intervention/within 7 days of hospital discharge
  Wechsler Adult Intelligence Scale-III Digit Span Test-Backward; number of correct trials, range: 0-14; higher scores indicate better performance
Cognitive function: executive function, working memory | Follow-up at 1 month post-hospital discharge
  Wechsler Adult Intelligence Scale-III Digit Span Test-Backward; number of correct trials, range: 0-14; higher scores indicate better performance
Cognitive function: executive function, working memory | Follow-up at 6 months post-hospital discharge
  Wechsler Adult Intelligence Scale-III Digit Span Test-Backward; number of correct trials, range: 0-14; higher scores indicate better performance
Cognitive function: executive function, working memory | Follow-up at 12 months post-hospital discharge
  Wechsler Adult Intelligence Scale-III Digit Span Test-Backward; number of correct trials, range: 0-14; higher scores indicate better performance
Cognitive function: executive function, set-shifting | Post-intervention/within 7 days of hospital discharge
  National Alzheimer's Coordinating Center Uniform Data Set: Oral Trail Making Test; time in seconds, range: 0-300; higher scores indicate worse performance
Cognitive function: executive function, set-shifting | Follow-up at 1 month post-hospital discharge
  National Alzheimer's Coordinating Center Uniform Data Set: Oral Trail Making Test; time in seconds, range: 0-300; higher scores indicate worse performance
Cognitive function: executive function, set-shifting | Follow-up at 6 months post-hospital discharge
  National Alzheimer's Coordinating Center Uniform Data Set: Oral Trail Making Test; time in seconds, range: 0-300; higher scores indicate worse performance
Cognitive function: executive function, set-shifting | Follow-up at 12 months post-hospital discharge
  National Alzheimer's Coordinating Center Uniform Data Set: Oral Trail Making Test; time in seconds, range: 0-300; higher scores indicate worse performance

CONTACTS AND LOCATIONS:
Overall Officials: Maya N Elias, PhD, MA, RN, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States